CLINICAL TRIAL: NCT00001920
Title: Investigation of Brain Function During Eyeblink Responding in Normal Volunteers and Patients With Schizophrenia (A Study of Behavior and Evoked Potentials)
Brief Title: Eye Blink Response in Healthy Volunteers and Adults With Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990166; 99-M-0166
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-02

CONDITIONS: Healthy; Schizophrenia
Keywords: Schizophrenia; Eyeblink; Evoked Potentials; Learning; Normal Volunteer; Healthy Volunteer
MeSH Terms: conditions — Schizophrenia

SUMMARY:
The purpose of this study is to explore how the brain works during particular memory tasks in people with schizophrenia and healthy volunteers.

Research has shown that patients with schizophrenia have structural and functional abnormalities in the hippocampus and cerebellum of their brains. These abnormalities are likely associated with the memory impairment experienced by these patients. Eye blink tests can provide information about memory acquisition involving the cerebellar and hippocampal regions. By altering the stimuli interval, these tests can distinguish between cerebellum-dependent memory associated with subliminal mnemonic encoding and hippocampus-dependent memory associated with conscious awareness. This study will use eyeblink tests to determine which type of memory is predominantly affected in schizophrenia.

Participants in this study will be screened with a physical and psychiatric examination. Participants will have an electroencephalogram (EEG), an electrocardiogram (ECG), and an electrodermal test. Evoked potentials and magnetic resonance imaging (MRI) scans of the brain may also be taken.

DETAILED DESCRIPTION:
Eyeblink conditioning is a paradigm that allows the study of aspects of the neural mechanism of memory in humans. This paradigm has been extensively studied in animals and human beings and its functional neuroanatomy appears to be well understood, involving the hippocampus and cerebellum. The performance on this task is most likely independent of subject motivation. Moreover, manipulation of the intervals between conditioned and unconditioned stimuli allows to study subliminal forms of mnemonic encoding ("delay" task) as well as learning that is associated with conscious awareness ("trace" task). This makes eyeblink conditioning particularly suited for study in patient populations, and particularly in schizophrenia where motivation and attention are frequently confounding factors in the study of memory processes.

Patients with schizophrenia have been reported to have hippocampal and possibly cerebellar structural and functional abnormalities, however eyeblink conditioning has been minimally studied in this patient population. We expect implicit forms of memory (cerebellum dependent) to be relatively spared as compared to declarative memory (hippocampus dependent) in schizophrenia.

We would like to test the hypothesis that patients with schizophrenia have deficits in acquiring the trace form of the task as opposed to the delay, where we assume they would be unimpaired as compared to normal controls. We would also like to study heart rate and skin conductance changes that occur during conditioning, since patients with schizophrenia have showed impaired autonomic function.

We also plan to study neurophysiological correlates of these behaviors with evoked response potentials (EP) and eventually functional magnetic resonance imaging (fMRI)

We expect EPs to show significant change in relation to development of the behavioral response. The association of awareness of the stimulus contingency with slow cortical potentials on the EEG will also be of interest.

ELIGIBILITY:
* INCLUSION CRITERIA

Controls:

No psychiatric or severe chronic medical illness at the time of the study, and by history. This includes the absence of substance abuse histories, learning disabilities and all DSM IV disorders. Medical histories will be evaluated by the investigators and medical conditions that are judged not to interfere with the study may be allowed.

No use of psychotropic substances in the last 3 months.

Age 18-60.

No family history of schizophrenia by subject report and possibly also by collateral report by at least one other family member.

Patients:

Schizophrenia, any subtype or schizoaffective disorder, depressed type by DSM IV (110).

Only concomitant medications should be neuroleptics and medications directed at controlling side effects (e.g. anticholinergics). An effort will be made to recruit patients on atypical neuroleptics, therefore attempting to minimize the anticholinergics, which might interfere with the acquisition of a conditioned response. When patients on anticholinergic treatment will be recruited as inpatients, a clinical evaluation of the risks and benefits of suspending anticholinergic treatment will be made and discussed with the patient. Anticholinergics will be withdrawn for a period equivalent to 3 half lives of the drug before attempting the study, if this is judged to be achievable with a relatively low risk and the patient agrees.

Age18-60.

EXCLUSION CRITERIA

Controls and Patients:

Impaired hearing.

Use of caffeine or tobacco in the 2 hours preceding the test.

Head trauma with loss of consciousness in the last year, or any evidence of functional impairment due to and persisting after head trauma.

All subjects who are unable to withstand the eyeblink testing will be excluded. Subjects who are not able to participate in the MRI (e.g. due to claustrophobia) will be studied to achieve a larger group for the behavioral experiments.

Subjects who are found to have eye lesions on exam.

Patients or healthy volunteers with a known risk from exposure to high magnetic fields (e.g. patients with pace makers) and those who have metallic implants (e.g. braces) in the head region (likely to create artifact on the MRI scans) will be excluded from participating in the MRI studies.

Patients:

Coexistence of another major mental illness at the time of the study. If the patients experienced other mental illnesses in the past (e.g. a learning disability or major depression), then this should be judged to be fully recovered.

Criteria for substance abuse met in the last 6 months.

Criteria for substance dependence met in the last year. If criteria for dependence were met in the past, then the duration of the disorder was less than 3 years, or not judged to have produced long term brain changes to allow the patient to be in the study.

Major concurrent medical illness likely to interfere with the acquisition of the task.

Concomitant medications which could interfere with performance on the task, excluding neuroleptics.

Presence of diskinetic movements of the face and tongue (likely to interfere with eyeblink measures, or of gross involuntary movements of the whole body (likely to interfere with positioning in the MRI scanner).

Pregnancy testing will be performed on women of childbearing age within the three days prior to MRI scanning.

Siblings of Patients with Schizophrenia:

The same inclusion criteria as normal volunteers, with the exception of family history, of course. In addition, the inclusion criteria for protocol #95-M-0150 will apply.

The same exclusion criteria as normal volunteers will apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 1999-08-30; Study Completion 2010-06-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Woodruff-Pak DS. Classical conditioning. Int Rev Neurobiol. 1997;41:341-66. doi: 10.1016/s0074-7742(08)60359-1. PMID 9378597
- [Background] Chen L, Bao S, Lockard JM, Kim JK, Thompson RF. Impaired classical eyeblink conditioning in cerebellar-lesioned and Purkinje cell degeneration (pcd) mutant mice. J Neurosci. 1996 Apr 15;16(8):2829-38. doi: 10.1523/JNEUROSCI.16-08-02829.1996. PMID 8786457
- [Background] Daum I, Schugens MM, Ackermann H, Lutzenberger W, Dichgans J, Birbaumer N. Classical conditioning after cerebellar lesions in humans. Behav Neurosci. 1993 Oct;107(5):748-56. doi: 10.1037//0735-7044.107.5.748. PMID 8280385